CLINICAL TRIAL: NCT02118519
Title: Use of Mesenchymal Stem Cells for the Repair of Articular Cartilage Disorder of Knee Using Intra-articular Injection of Mesenchymal Cells Alone or Mesenchymal Cells With Platelet Lysate
Brief Title: Mesenchymal Stem Cells in Knee Cartilage Injuries
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Fatima Jamali, Researcher, University of Jordan
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KneeUJCTC
Record Dates: First submitted 2014-01-24; First posted 2014-04-21 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Articular Cartilage Disorder of Knee; Osteoarthritis, Knee
Keywords: Bone marrow derived Mesenchymal Stem Cells; Knee articular cartilage injury; Chondrogenesis; orthopedics
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- mesenchymal stem cells (Active Comparator): Autologous Mesenchymal Stem Cells primed prior to intra articular injection into knees of patients with advanced articular cartilage injury
  Interventions: Biological: Autologous Mesenchymal Stem Cells
- mesenchymal cells&platelet lysate (Active Comparator): Autologous Mesenchymal Stem Cells primed prior to intra articular injection with platelet lysate into knees of patients with advanced articular cartilage injury
  Interventions: Biological: Autologous Mesenchymal Stem Cells

INTERVENTIONS:
Biological: Autologous Mesenchymal Stem Cells — Comparison of clinical outcomes of patients injected by mesenchymal stem cells only with patients injected with mesenchymal stem cells supported by platelet lysate

SUMMARY:
Induction of autologous repair chondrogenesis to regenerate injured articular cartilage using bone marrow mesenchymal stem cells (MSCs) after in vitro expansion under restricted culturing conditions.

DETAILED DESCRIPTION:
Fourteen patients from both genders, age range 40-68, will be enrolled according to strict inclusion and exclusion criteria, divided into two equal groups based upon receiving autologous MSCs alone, or MSCs supported by platelet lysate through percutaneous injection.

The patients are followed by clinical assessment, laboratory investigations as well as magnetic resonance imaging (MRI) of the injected knee.

The investigators hypothesize that the two groups will give satisfactory clinical outcomes, but the investigators are looking forward to assessing the best product that will activate chondrogenesis and heal cartilaginous injury.

ELIGIBILITY:
Inclusion Criteria:

* MRI must show moderate/severe articular injury
* Serum collagen II must be above the normal value.
* Lesion site: Femoral and Tibial condyles or patella
* Admission of steroid , NSAID, pain killers must be stopped before 1 month

Exclusion Criteria:

* Lesion size
* PT and PTT not within normal value
* Complete blood count ( Hb, PCV, and RBC) not within the normal value
* HIV and Hepatitis Antigens (B and C) detection

Ages: 40 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Assessing the therapeutic benefits of the injected Autologous Mesenchymal Stem Cells. | 12 months

SECONDARY OUTCOMES:
Assessment of the articular cartilage healing in osteoarthritic patients through intra articular injection of Autologus Mesenchymal stem cell with/or without supported product. | 12 months
  For every patient tests would be performed repeated at 6, and 12 months post-injection.

CONTACTS AND LOCATIONS:
Overall Officials: Abdallah Awidi, MD, Study Director — Cell Therapy Center; Mahasen S Najjar, MD, Principal Investigator — Jordan University Hospital; Hiba Khalil, PhD, Principal Investigator — Al-Neelain University
Locations (1):
- Cell Therapy Center, Jordan University Hospital, Amman, Jordan

REFERENCES:
- [Derived] Al-Najar M, Khalil H, Al-Ajlouni J, Al-Antary E, Hamdan M, Rahmeh R, Alhattab D, Samara O, Yasin M, Abdullah AA, Al-Jabbari E, Hmaid D, Jafar H, Awidi A. Intra-articular injection of expanded autologous bone marrow mesenchymal cells in moderate and severe knee osteoarthritis is safe: a phase I/II study. J Orthop Surg Res. 2017 Dec 12;12(1):190. doi: 10.1186/s13018-017-0689-6. PMID 29233163